CLINICAL TRIAL: NCT01690546
Title: An Open Label, Flexible Dose Study of Very Low Doses of Naltrexone-Buprenorphine Transfer to Extend-Release Naltrexone (VIVITROL®) in Opioid Addiction
Brief Title: Low Dose Naltrexone-buprenorphine Transfer to Vivitrol Injection in Opioid Dependence
Acronym: BUP/NXT-VIVI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Paolo Mannelli (Other)
Collaborators: Alkermes, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Paolo Mannelli, Associate Professor of Psychiatry, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00036909
Record Dates: First submitted 2012-09-19; First posted 2012-09-21 (Estimated); Results first posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-04

CONDITIONS: Opiate Dependence
Keywords: Opioid Addiction; Addiction; Drug Dependence
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive; Substance-Related Disorders | interventions — Naltrexone; vivitrol; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BUP/VLNXT to VIVITROL (Experimental): On days 1-3, participants will receive buprenorphine/naloxone daily, starting at a dose of 4 mg, progressively decreasing to 2 mg on Days 2-3 and very low dose naltrexone at 0.25 mg to 1 mg on Days 1-3, 2 to 6 mg on Day 4 and 10 mg to 50 mg on Days 5-7. VIVITROL injection will be administered on Day 8 at 380 mg.
  Interventions: Drug: very low dose naltrexone; Drug: extended release naltrexone; Drug: buprenorphine/naloxone

INTERVENTIONS:
Drug: very low dose naltrexone — On days 1-3, participants will receive buprenorphine/naloxone daily, starting at a dose of 4 mg, progressively decreasing to 2 mg on Days 2-3 and very low dose naltrexone at 0.25 mg to 1 mg on Days 1-3, 2 to 6 mg on Day 4 and 10 mg to 50 mg on Days 5-7. VIVITROL injection will be administered on Day 8 at 380 mg.
Drug: extended release naltrexone — On days 1-3, participants will receive buprenorphine/naloxone daily, starting at a dose of 4 mg, progressively decreasing to 2 mg on Days 2-3 and very low dose naltrexone at 0.25 mg to 1 mg on Days 1-3, 2 to 6 mg on Day 4 and 10 mg to 50 mg on Days 5-7. VIVITROL injection will be administered on Day 8 at 380 mg.
  Other Names: Vivitrol
Drug: buprenorphine/naloxone — On days 1-3, participants will receive buprenorphine/naloxone daily, starting at a dose of 4 mg, progressively decreasing to 2 mg on Days 2-3 and very low dose naltrexone at 0.25 mg to 1 mg on Days 1-3, 2 to 6 mg on Day 4 and 10 mg to 50 mg on Days 5-7. VIVITROL injection will be administered on Day 8 at 380 mg.
  Other Names: Suboxone

SUMMARY:
The purpose of this study is to evaluate a very low dose naltrexone-buprenorphine treatment to transfer opioid dependent individuals to extended release naltrexone injection (Vivitrol). The hypothesis is that patients will complete the transfer to Vivitrol successfully, finding the treatment acceptable and showing minimal withdrawal discomfort.

DETAILED DESCRIPTION:
Thirty-five opioid dependent (OD) volunteers seeking treatment will be enrolled in an open-label, flexible-dosing, outpatient trial at Duke Addictions Program. On days 1-3, participants will receive buprenorphine/naloxone daily at a starting dose of 4mg, progressively decreasing to 2 mg on days 2- 3. Participants will also receive very low dose naltrexone (VLNTX) at a dose of 0.25 mg to 1mg on Days 1-3, 2 to 6 mg on Day 4 and between 10 and 50 mg on Days 5-7. Then a VIVITROL injection, 380 mg, will be administered on Day 8.

Evaluations will occur daily for up to 6 hours until 1 day after VIVITROL injection and then weekly for 4 weeks. Patients will receive ancillary medications as needed and weekly psychosocial intervention. At the end of the study, participants will be offered outpatient treatment of OD at the study site, or will be referred to other treatment programs.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18 to 65 years of age who meet DSM-IV criteria for OD of at least six months duration, supported by a positive urine for opiates and a positive naloxone challenge test if the diagnosis is unclear.
2. Individuals must be capable of giving informed consent and capable of complying with study procedures.
3. Participants will be asked to provide locator information including the address and telephone number of a non-drug abusing relative or friend who can reach the participant in emergencies.

Exclusion Criteria:

1. Individuals currently prescribed or regularly taking opiates for chronic pain or medical illness.
2. Individuals regularly using licit or illicit methadone or BUP.
3. Individuals meeting DSM-IV criteria for schizophrenia, schizoaffective or psychotic disorders, or psychiatric disorder (other than substance abuse) requiring intervention.
4. Individuals who are medically unstable, or have liver enzyme function tests greater than two times normal.
5. Individuals with current suicidal risk or 1 or more suicide attempts within the past year.
6. History of accidental drug overdose in the last three years or any other significant history of overdose following detoxification, defined as an episode of opioid-induced unconsciousness or incapacitation.
7. Nursing/pregnant women, or failure in a sexually active man or woman to use adequate contraceptive methods (e.g., oral or depot contraceptives, foam, sponges, and/or condoms)
8. Individuals who are dependent on any other drugs (excluding nicotine)
9. Individuals with known sensitivity to BUP, VIVITROL, NTX, naloxone.
10. Individuals who are court-mandated to treatment.
11. Individuals who have a current or pending legal status, or any other condition that would make them unlikely to be available for the duration of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Mannelli, MD, Principal Investigator — Duke University Health Systems
Locations (1):
- Duke University Medical Center / Civitan Building, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 participants signed consent. 3 participants were screen failures. 35 participants started study.
Period: Overall Study
Arm/Group | BUP/VLNXT to VIVITROL
Started | 35
Extended Release Injectable NTX | 27
Completed | 26
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | BUP/VLNXT to VIVITROL
Number analyzed (Participants) | 35
Age, Continuous [Mean (Full Range); unit: years] | 40.1 [25 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 26
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 26
  Caucasian | 9
Years of Opioid use [Mean (Full Range); unit: years] | 9.7 [7 to 18]

OUTCOME MEASURES:

1. Primary Outcome: Retention in Treatment
Description: After the initial titration period for opioid withdrawal (of up to 8 days), patients will receive the Vivitrol injection. Then, we will follow patients for retention out to 4 weeks.
Time Frame: 4 weeks
Population: All participants who received the Extended Release Injectable NTX
Measure: Number; unit: participants
Arm/Group | BUP/VLNXT to VIVITROL
Number analyzed (Participants) | 27
participants | 26

2. Secondary Outcome: Withdrawal Intensity as Measured by the Clinical Opiate Withdrawal Scale (COWS)
Description: After the initial titration period for opioid withdrawal (of up to 8 days), patients will receive the Vivitrol injection. Then, we will follow patients for retention out to 4 weeks and record the total time they remained in treatment.
  COWS rates eleven common opiate withdrawal signs or symptoms. The summed scores ranged from 0-48, with 5-12 = mild; 13-24 = moderate; 25-36 = moderately severe; more than 36 = severe withdrawal.
Time Frame: 4 weeks
Population: All participants who received the Extended Release Injectable NTX
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BUP/VLNXT to VIVITROL
Number analyzed (Participants) | 27
units on a scale | 0.64 (1.29)

3. Secondary Outcome: Withdrawal Intensity as Measured by the Subjective Opiate Withdrawal Scale (SOWS)
Description: After the initial titration period for opioid withdrawal (of up to 8 days), patients will receive the Vivitrol injection. Then, we will follow patients for retention out to 4 weeks and record the total time they remained in treatment.
  SOWS contains 16 symptoms whose intensity the patient rates on a scale of 0 (not at all) to 4 (extremely). Total score range is 0 - 64; the higher the score the more withdrawal symptoms.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BUP/VLNXT to VIVITROL
Number analyzed (Participants) | 27
units on a scale | 1.52 (3.19)

4. Secondary Outcome: Craving
Description: Craving, assessed with a 100-point Visual Analog Scale (VAS), ranging from 'not at all' (0) to 'more than ever' (100). The higher the score the higher the craving.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BUP/VLNXT to VIVITROL
Number analyzed (Participants) | 27
units on a scale | 5.12 (14.41)

5. Secondary Outcome: Illicit Drug Use, Measured by Urine Drug Testing
Description: number of participants that tested positive for marijuana, cocaine, and opiates.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | BUP/VLNXT to VIVITROL
Number analyzed (Participants) | 26
participants
  Marijuana | 11
  Cocaine | 3
  Opiates | 4

6. Secondary Outcome: Satisfaction With Treatment, Measured by a Treatment Satisfaction Questionnaire
Description: Questionnaire consisted of 3 questions.
  1. Were you satisfied with the treatment (range 1-5): Completely satisfied (1) to completely dissatisfied (5).
  2. Were you satisfied with withdrawal treatment (range 1-5): Minimal withdrawal (1) to worse than ever (5).
  3. Did the medication help (range 1-5): Helped a lot (1) to No it did not help (5).
  Lower scores represent greater satisfaction.
Time Frame: Day 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BUP/VLNXT to VIVITROL
Number analyzed (Participants) | 27
units on a scale
  Were you satisfied with the treatment | 1.31 (0.84)
  Were you satisfied with withdrawal treatment | 2.04 (0.82)
  Did the medication help | 1.69 (0.93)

7. Secondary Outcome: Percentage of Participants Who Adhered to Study Visits.
Time Frame: baseline to end of study (approximately 40 days)
Measure: Number; unit: percentage of participants
Arm/Group | BUP/VLNXT to VIVITROL
Number analyzed (Participants) | 35
percentage of participants | 74

8. Secondary Outcome: Percentage of Participants With Adherence to Medication (Naltrexone)
Description: Participant who took Naltrexone as prescribed.
Time Frame: Day 1 to Day 8 (+/- 2 days)
Measure: Number; unit: percentage of participants
Arm/Group | BUP/VLNXT to VIVITROL
Number analyzed (Participants) | 35
percentage of participants | 100

9. Secondary Outcome: Use of Ancillary Medications.
Description: Number of participants that took ancillary medication
Time Frame: baseline to week 1
Measure: Number; unit: participants
Arm/Group | BUP/VLNXT to VIVITROL
Number analyzed (Participants) | 35
participants | 35

10. Secondary Outcome: Number of Participants That Self Reported Illicit Drug Use
Description: Participants reported on any illicit drug use to include Cocaine marijuana opiates
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | BUP/VLNXT to VIVITROL
Number analyzed (Participants) | 26
participants
  Marijuana | 10
  Cocaine | 3
  Opiates | 4

ADVERSE EVENTS:
Arm/Group | BUP/VLNXT to VIVITROL
Serious Adverse Events (participants affected / at risk) | 1/35
Other Adverse Events (participants affected / at risk) | 6/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BUP/VLNXT to VIVITROL (N=35)
persecutory ideations (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BUP/VLNXT to VIVITROL (N=35)
Increased Withdrawal Symptoms (General disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No